CLINICAL TRIAL: NCT05909449
Title: Improving Posture and Health-Related Physical Fitness Parameters of Primary Care Providers to Individuals With Disabilities
Brief Title: Improving Posture Parameters of Primary Care Providers to Individuals With Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gulser CINBAZ, Research Asistant, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-9169
Record Dates: First submitted 2023-05-10; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-04

CONDITIONS: Physical Disability
Keywords: posture; Physical Fitness; care provider
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research group (Experimental): provide primary care services to individuals with physical disabilities
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — participants will be given a structured home exercise program

SUMMARY:
The aim of this research is to create and implement an exercise program so that primary caregivers can have the correct posture and improve health-related physical fitness parameters.

DETAILED DESCRIPTION:
It is planned to include at least 40 volunteers between the ages of 18-65 who meet the inclusion criteria and provide primary care services to individuals with disabilities who attend Sportive Skills and Coordination Training Centers operating in the provinces of Istanbul and Gaziantep within the body of the Foundation for the Physically Disabled. Musculoskeletal complaints of caregivers related to the care process (neck pain, low back pain and upper extremity pain), physical fitness parameters (functional capacity and shortness-flexibility, balance and footpad pressure distribution), the effects of the caregiving process on the caregiver and mental well-being will be evaluated.

After the first evaluation, the participants will be given an informative training seminar on the effects of exercise on healthy life and the regulation of ergonomics in our behaviors. After the seminar, participants will be included in a structured home exercise program. The home exercise program prepared by the research team and recorded on video will be delivered to the participants. The exercise program will be continued for 6 weeks, 3 days a week. The exercise program will be prepared weekly to advance to the next level. Exercise compliance and attendance will be monitored weekly by the researchers. Evaluations will be repeated at the end of the 6-week exercise program.

Establishment of an exercise program: In the light of the data obtained as a result of the evaluations, an individual-specific exercise program will be created. The exercises will be taught one-on-one to the participants. With the exercise video prepared by the project team and sent to the patients, the participants will be prevented from forgetting the exercises and they will be stimulated to do the exercises correctly. The content of the exercise program will include exercises that include aerobic, strengthening and flexibility components. The exercise program will take approximately 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65
* To give primary care to a person with a physical disability
* Being caring for at least 6 months
* Voluntarily performing care
* Being able to understand and read Turkish as a language
* To have sufficient cognitive level to answer the scale questions with the basic interview
* Volunteer to participate in and maintain an exercise program
* Regularly participating in the evaluation and exercise program defined during the project process

Exclusion Criteria:

* Caring for a paid job other than voluntarily
* Encountering a disease related to the caregiver during the working process
* Having any known musculoskeletal disease
* Having a known spinal problem such as scoliosis, kyphosis, kyphoscoliosis
* Having undergone surgery affecting the musculoskeletal system in the last 1 month
* History of uncontrollable arrhythmia and/or hypertension
* Having any neurological, cardiovascular, respiratory, orthopedic and metabolic disease that will prevent participation in the exercise program
* Being pregnant for female individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-07-03 (Estimated)

PRIMARY OUTCOMES:
The Nordic Musculoskeletal Questionnaire | twice (before and after 6 week exercise program)
  NMQ is a questionnaire that evaluates low back, neck, shoulder and general musculoskeletal complaints with standardized questions. In NMQ; Pain and discomfort in nine mapped and marked areas of the body (feet-ankles, knees, thighs-hips, wrists-hands, waist, elbows, back, shoulders, neck), and whether this is interfering with normal work being questioned
Oswestry Low Back Pain Disability Index | twice (before and after 6 week exercise program)
  It consists of 10 titles (Pain sensitivity, self-care, weight lifting, reading, headaches, concentration, study/work, driving, sleep, and social activities). Each question has 6 answer options that measure the severity of pain or limitation. Scoring is done between 0-5. The total score is between 0-50. There is no limitation between 0-4 points according to the total score; 5-14 mild limitation; 15-24 moderately restricted; 25-34 severe limitation; 34 and above are classified as completely restricted
The shortened disabilities of the arm, shoulder and hand questionnaire (Quick DASH) | twice (before and after 6 week exercise program)
  Q-DASH is a regional outcome measure developed for upper extremity musculoskeletal disorders and includes 11 questions. Each question is scored on a 5-point scale and a final score ranging from 0 (no disability) to 100 (severe disability) is calculated.
The Oswestry Disability Index (ODI) | twice (before and after 6 week exercise program)
  It consists of a total of 10 items measuring the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleeping, traveling and the degree of pain. Each item is graded between 0-5. The maximum score is 50 points; It is evaluated as severe disability between 31-50 points, moderate between 11-30 points and mild disability between 1-10 points.
Two Minute Walk Test (2MWT) | twice (before and after 6 week exercise program)
  2DYT is carried out in a 30 meter long corridor. The starting and ending points are determined by marking the corridor every 3 meters. A colored cone is placed in the turning zones. Participants are asked to walk the 30-meter corridor for 2 minutes at their own walking speed without running. Distance traveled in 2 minutes is recorded
Sit and Reach Test | twice (before and after 6 week exercise program)
  The test will be used to assess lower extremity flexibility. For this test, the participants will be asked to rest their feet on the test bench while in a long sitting position with their knees straight, and without bending their knees, put their hands on each other and extend their arms towards the test bench in front. 3 repetitions will be made and the average value will be recorded.
force platform | twice (before and after 6 week exercise program)
  Balance and sole pressure distribution will be evaluated with the force platform. Balance parameters and footpad pressure distribution evaluations of the cases will be recorded with a force platform (Matscan, TekScan, Boston, MA, USA) with a recording speed of 100Hz and a resolution of 4 senses/cm². Measurements; It will be performed with eyes open and closed, in free standing position and on one foot (first on the dominant, then on the non-dominant foot). For the measurement at each position, force platform records will be taken for 30 seconds. Analysis of the data will be done using Matscan 7.10 (TekScan, Boston, MA) software provided by the manufacturer. To evaluate the balance, center of gravity range of motion (cm2), antero-postero oscillation (cm) and medio-lateral oscillation (cm) values will be recorded.
Back reach test | twice (before and after 6 week exercise program)
  This test evaluates shoulder flexibility. While in a standing position, one arm is externally rotated with the fingers extended and the palm facing the back, reaching the lowest point of the back over the shoulder towards the back and while doing this, the other arm is internally rotated, with the palm facing forward and the fingers again. While in extension, he will be asked to reach the highest point on his back. The distance between the middle fingers placed on the back will be recorded
The Zarit Care Burden Scale (ZBVYS) | twice (before and after 6 week exercise program)
  It was developed by Zarit et al to evaluate the effects of the caregiving process on the caregiver. It consists of 22 statements that determine the effect of caregiving on the life of the individual. Although a maximum of 88 points can be obtained from a 5-point Likert-type scale (1=never, 5=always), higher scores indicate higher caregiving burden
Warwick-Edinburgh Mental Well-being | twice (before and after 6 week exercise program)
  It was developed by Tennant et al. to measure the mental well-being of the caregiver. The scale consists of 14 items covering psychological well-being and subjective well-being. It is a 5-point Likert-type scale, with the lowest 14 points and the highest 70 points. High scores from the scale indicate high mental (psychological) well-being.

CONTACTS AND LOCATIONS:
Overall Officials: NİLÜFER KABLAN, Study Director — associate professor
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No